CLINICAL TRIAL: NCT02237950
Title: A Phase 3, Double-blind, Multicentre, Randomised, Placebo-controlled Study to Determine the Efficacy and Safety of SPL7013 Gel to Prevent the Recurrence of Bacterial Vaginosis
Brief Title: Efficacy and Safety Study of SPL7013 Gel to Prevent the Recurrence of Bacterial Vaginosis (BV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Starpharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPL7013-017
Record Dates: First submitted 2014-09-05; First posted 2014-09-12 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole; astodrimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1% SPL7013 Gel (Experimental): Inserted in to the vagina on alternate days (i.e. every other day) for 16 weeks
  Interventions: Drug: Metronidazole oral tablets 500mg; Drug: 1% SPL7013 Gel
- Placebo Gel (Placebo Comparator): Inserted in to the vagina on alternate days (i.e. every other day) for 16 weeks
  Interventions: Drug: Metronidazole oral tablets 500mg; Drug: Placebo gel

INTERVENTIONS:
Drug: Metronidazole oral tablets 500mg — One tablet taken orally twice daily for seven consecutive days
Drug: 1% SPL7013 Gel — 5g inserted in to the vaginal on alternate days (i.e. every other day) for 16 consecutive weeks.
  Other Names: VivaGel; astodimer sodium
  Arms: 1% SPL7013 Gel
Drug: Placebo gel — 5g inserted in to the vagina on alternate days (i.e. every other day) for 16 consecutive weeks
  Arms: Placebo Gel

SUMMARY:
A double-blind, phase 3 study to determine the efficacy of SPL7013 Gel when administered on alternate days for 16 weeks, compared to placebo gel in preventing the recurrence of BV in women with a history of recurrent BV.

DETAILED DESCRIPTION:
Eligible participants, with both a history of recurrent BV and a current episode of BV, will receive a seven-day course of oral metronidazole. Participants who are successfully treated for their BV, and continue to be eligible, will be randomly assigned to receive either 1% SPL7013 Gel or placebo gel on alternate days at bed-time for 16 consecutive weeks.

The primary endpoint will be determined at the conclusion of this 16 week treatment phase.

Participants who experience a BV recurrence will be considered to have completed the study. Such participants will receive BV treatment in line with local practice and will not attend any further study visits.

Participants who successfully reach Week 16 without a BV recurrence will enter a 12-week follow-up phase to Week 28.

Participants will attend a study visit at 4-weekly intervals throughout the duration of the study to Week 28 (or up to the point of BV recurrence) to assess recurrence of BV and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Current active episode of BV (diagnosis defined as: At least 3 of the 4 Amsel criteria; Nugent score of at least 4; presence of BV-related symptoms)
* History of recurrent BV (at least 3 episodes in previous year including current episode)
* Using an effective method of contraception

Exclusion Criteria:

* Test positive for a sexually transmitted infection
* Presence of genital Herpes Simplex Virus (HSV) lesions or Human Papilloma Virus (HPV) lesions requiring treatment
* Abnormal pelvic exam, including presence of other vaginal or urinary tract infections
* Pregnancy

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 586 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Paull, PhD., Study Chair — Starpharma Pty Ltd
Locations (45):
- United States (37):
  - University of Alabama, Birmingham, Alabama
  - Montgomery Women's Health Associates, Montgomery, Alabama
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Precision Research Institute, San Diego, California
  - Women's Health Care, San Diego, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Downtown Women's Health Care, Denver, Colorado
  - The Community Research South Florida, Hialeah, Florida
  - Florida Medical Center and Research Inc., Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Community Medical Research, Miami Beach, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Atlanta Medical Research Institute, Alpharetta, Georgia
  - Urban Family Practice Associates, Marietta, Georgia
  - Heartland Research Associates, LLC, Newton, Kansas
  - Women's Healthcare Specialists, Paw Paw, Michigan
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Alegent Creighton Health, Omaha, Nebraska
  - Affiliated Clinical Research, Las Vegas, Nevada
  - Lawrence OB-GYN Associates, Lawrenceville, New Jersey
  - PMG Research of Cary, LLC, Cary, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Radiant Research, Akron, Ohio
  - Radiant Research, Columbus, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Clinical Research Advantage, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Women's Physician Group, Memphis, Tennessee
  - Practice Research Organization, Dallas, Texas
  - Radiant Research, San Antonio, Texas
  - Jordan River Family Medicine, South Jordan, Utah
  - Clinical Trials of Virginia, Richmond, Virginia
  - Women's Clinical Research Center, Seattle, Washington
- Canada (5):
  - Medicine Professional Corporation, Kitchener, Ontario
  - SKDS Research Inc, Newmarket, Ontario
  - Healthy Image Centre, Windsor, Ontario
  - DIEX Recherche Montreal Inc, Montreal, Quebec
  - DIEX Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Puerto Rico (3):
  - Torre Auxillo Mutuo, Hato Rey
  - Latin Clinical Trial Center, San Juan
  - University of Puerto Rico, San Juan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Started | 295 | 291
Completed | 247 | 243
Not Completed | 48 | 48

BASELINE CHARACTERISTICS:
Population: Analysis population is the modified intent-to-treat analysis population. One patient was excluded compared with the intent-to-treat population because they were dispensed medication but returned all unused.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% SPL7013 Gel | Placebo Gel | Total
Number analyzed (Participants) | 294 | 291 | 585
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (7.23) | 31.6 (6.99) | 31.6 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 294 | 291 | 585
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of BV Where a Diagnosis of BV is Defined as the Presence of at Least 3 Clinical Findings
Description: Number of participants with a recurrence of BV, where a diagnosis of BV is defined as the presence of at least 3 clinical findings (Amsel criteria)
Time Frame: At or by the Week 16 visit
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 294 | 291
Participants | 130 | 158
Statistical Analysis 1: Comparison: 1% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.015, Regression, Logistic

2. Secondary Outcome: Time to Recurrence of BV Where a Diagnosis of BV is Defined as the Presence of at Least 3 Clinical Findings
Description: Time to recurrence of BV (days), where a diagnosis of BV is defined as the presence of at least 3 clinical findings (Amsel criteria)
Time Frame: At or by the Week 16 visit
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 294 | 291
days | 105 [98 to 111] | 99 [87 to 106]
Statistical Analysis 1: Comparison: 1% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.007, Log Rank

3. Secondary Outcome: Recurrence of Patient-reported BV Symptoms
Description: Number of participants with self-reported BV symptoms (vaginal discharge and/or odor)
Time Frame: At or by the Week 16 visit
Population: Modified Intent-to-Treat, excluding patients with missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 269 | 266
Participants | 75 | 108
Statistical Analysis 1: Comparison: 1% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.002, Regression, Logistic

4. Secondary Outcome: Recurrence of Individual Amsel Criteria
Description: Number of participants with positive individual Amsel criterion
  - Clue cells representing at least 20% of total epithelial cells
Time Frame: At or by the Week 16 visit
Population: Modified Intent-to-Treat, excluding patients with missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 274 | 273
Participants | 104 | 132
Statistical Analysis 1: Comparison: 1% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.014, Regression, Logistic

5. Secondary Outcome: Recurrence of BV as Determined by Presence of a Nugent Score of 7-10
Description: Number of participants with a recurrence of BV as determined by presence of a Nugent score of 7-10 (BV), where 0-3 is normal, and 4-6 is intermediate.
Time Frame: At or by the Week 16 visit
Population: Modified Intent-to-Treat, excluding patients with missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 247 | 273
Participants | 95 | 135
Statistical Analysis 1: Comparison: 1% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.012, Regression, Logistic

6. Secondary Outcome: Recurrence of BV Where a Diagnosis of BV is Defined as the Presence of at Least 3 Clinical Findings
Description: as for outcome 1
Time Frame: At or by the Week 24 visit
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 294 | 291
Participants | 194 | 213
Statistical Analysis 1: Comparison: 1% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.059, Regression, Logistic

7. Secondary Outcome: Recurrence of BV According to the Composite Definition of at Least 3 Clinical Findings (Amsel Criteria) and a Nugent Score of 4-10.
Description: Number of participants with a recurrence of BV according to the composite definition of at least 3 clinical findings (Amsel criteria) and a Nugent score of 4-10 (intermediate to BV), where 0-3 is normal.
Time Frame: At or by the Week 16 visit
Population: Modified Intent-to-Treat, excluding patients with missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 276 | 276
Participants | 81 | 111
Statistical Analysis 1: Comparison: 1% SPL7013 Gel vs Placebo Gel; Test type: Superiority; p = 0.008, Regression, Logistic

8. Secondary Outcome: Change From Baseline in Brief Index of Sexual Functioning for Women Questionnaire Composite Score
Description: Change from baseline in brief index of sexual functioning for women (BISF-W) questionnaire composite score. The composite score includes scores from dimensions (D) of thoughts/desire (D1, 0-12), arousal (D2, 0-12), frequency of sexual activity (D3, 0-12), receptivity/initiation (D4, 0-12), pleasure (D5, 0-12), relationship satisfaction (D6, 0-12), and any problems affecting sexual functioning (D7, 0-16). The composite score is calculated as D1+D2+D3+D4+D5+D6-D7 with a range of -16 to +75. A positive change in composite score from baseline to Week 16 reflects an improvement in sexual functioning, with a greater change in score indicating a greater improvement in sexual functioning.
Time Frame: Baseline to Week 16
Population: Analysis population includes only those participants who completed the survey, which was optional.
Measure: Mean (95% Confidence Interval); unit: change in score on a scale
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 163 | 166
change in score on a scale | 1.6 [-0.5 to 3.7] | 0.1 [-2.0 to 2.1]

9. Secondary Outcome: Adverse Events (AEs)
Description: Number of participants with genitourinary AEs considered potentially related to study treatment
Time Frame: From Baseline to end of Week 28
Population: Safety population was all patients in the Intent-to-Treat population, but excluding those who later returned all the study medication unused.
Measure: Count of Participants; unit: Participants
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Number analyzed (Participants) | 294 | 291
Participants | 37 | 33

ADVERSE EVENTS:
Description: Safety population was all patients in the Intent-to-Treat population, but excluding those who later returned all the study medication unused.
Arm/Group | 1% SPL7013 Gel | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 4/294 | 3/291
Other Adverse Events (participants affected / at risk) | 92/294 | 80/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% SPL7013 Gel (N=294) | Placebo Gel (N=291)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Hemiplegic migraine (Nervous system disorders) | 0 (0) | 1 (1)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1% SPL7013 Gel (N=294) | Placebo Gel (N=291)
Nasopharyngitis (Infections and infestations) | 9 | 15
UTI (Infections and infestations) | 28 | 10
Vulvovaginal candidiasis (Infections and infestations) | 47 | 35
Vulvovaginal mycotic infection (Infections and infestations) | 14 | 16
Headache (Nervous system disorders) | 17 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, PIs can publish data only after study data are published collectively.